CLINICAL TRIAL: NCT05306743
Title: Pragmatic Evaluation of a Quality Improvement Program for People Living With Modifiable High-risk COPD (PREVAIL)
Brief Title: PRagmatic EVAluation of a Quality Improvement Program for People Living With Modifiable High-risk COPD.
Acronym: PREVAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Observational and Pragmatic Research Institute (Other)
Collaborators: The DARTNet Institute (DI) (Unknown); AstraZeneca (Industry); Optimum Patient Care Global Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OPRI-2003
Record Dates: First submitted 2022-03-13; First posted 2022-04-01 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Airway Disease; Quality Improvement Program
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A total of 126 primary care teams (PCT) will be enrolled in the trial; 63 PCTs will be randomized to the intervention arm and receive the CONQUEST QIP, and 63 to the control arm where they will receive care as usual.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONQUEST Intervention Arm (Experimental): Intervention arm clusters will receive the CONQUEST quality improvement program.
  Interventions: Other: CONQUEST Quality Improvement Program
- Delayed Intervention Arm (Other): The CONQUEST quality improvement program will be rolled-out to the delayed intervention practices at the end of the outcome evaluation period.
  Interventions: Other: CONQUEST Quality Improvement Program

INTERVENTIONS:
Other: CONQUEST Quality Improvement Program — CONQUEST supports primary healthcare professionals to diagnose, assess, and optimize the management of their patients with modifiable high-risk COPD, through the promotion of guideline-based care. CONQUEST will promote management according to four "Quality Standards" for the care of modifiable high-risk COPD patients. The Quality Standards can be summarized as the timely and appropriate: Identification of high-risk patient groups for assessment; Assessment of disease and quantification of future risk; Non-pharmacological and pharmacological intervention; Follow-up. CONQUEST program will promote adherence to these standards through the use of electronic medical record -based algorithms for the identification of high-risk patients and clinical decision support resources. All decisions regarding patient management are made entirely at the discretion of the clinicians and patients who together negotiate the preferred course of action during consultations.

SUMMARY:
A 3-year cluster randomized controlled trial of the impact of a quality improvement and clinical decision support package versus usual care for patients with modifiable high-risk chronic obstructive pulmonary disease with or without a current diagnosis.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a frequently underdiagnosed major health problem, responsible for over 250 million cases of disease and 3 million deaths (5% of all deaths) worldwide in 2015. Despite resulting in more than $30 billion in direct healthcare costs in the USA, and causing significant morbidity and lost days of work, COPD remains a globally under-recognised condition, with an estimated 60% of cases undetected at any one time, and frequently misdiagnosed in smokers and people with asthma.

Even once diagnosed, about two thirds of patients will have already experienced significant lung function decline or previous serious exacerbations, indicating that opportunities for earlier diagnosis may have been lost. The consequences of this have been summarized persuasively using data from large population-based studies of patients, demonstrating higher future risk of exacerbations, accelerated lung function decline, greater risk of cardiovascular events, higher mortality rates, and larger healthcare costs in late diagnosed patients with a symptomatic history.

Several proof of principle studies have demonstrated the feasibility of case finding in primary care, however, in practice it is patchily implemented if at all, with inconsistent evidence demonstrating significant positive impact. This is partially because post-case finding, patient follow-up and management can be poor and significant subgroups of COPD patients with frequent exacerbations or high symptom scores remain undertreated or under-monitored according to quality standards. Such patients represent a high-risk "phenotype" in whom risk may be reduced with dedicated measures taken for individualized, targeted management. This may be achieved by analyzing patient electronic medical records (EMR) data as a means to identify patients with modifiable, high-risk COPD in whom there remains options to further optimize their treatment according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) recommendations.

The CONQUEST intervention (Collaboration on a Quality Improvement Initiative to Achieve Excellence in Standards of COPD Care) will address areas for optimization of the management of patients with modifiable high-risk COPD, or potential COPD, through a targeted Quality Improvement Program (QIP) in primary care practices. The intervention will implement validated algorithms (appropriately adapted for CONQUEST) to identify patients with modifiable high-risk COPD or undiagnosed patients with potential modifiable high-risk COPD, and support their management through a multicomponent package incorporating Clinical Decision Support (CDS).

Parallel to this, the pragmatic cluster randomized controlled trial - "PREVAIL" (PRagmatic EVAluation of a quality Improvement program for people Living with modifiable high-risk COPD) will be conducted evaluating the effectiveness of the CONQUEST intervention compared to usual care. Primary care teams will be the cluster unit of randomization.

Because of the established relationship between risk of major cardiac events and exacerbations, the effectiveness of the CONQUEST program will be evaluated in terms of COPD exacerbations and cardiovascular or respiratory events. The design of this trial presents a unique opportunity to compare major adverse cardiac or respiratory events (MACRE) outcomes in a naturally-occurring group of patients who are both frequent exacerbators and either treatment-naïve or undertreated at trial baseline, and to measure these outcomes over a period of time comparatively longer than the standard 52 weeks of many clinical trials of COPD medications.

ELIGIBILITY:
As a cluster randomized controlled trial, participants in PREVAIL are the Primary Care Teams. The PREVAIL CRT adopts the definition of PCT from the Agency for Healthcare Research and Quality, "a group of primary care practice personnel who identify as members of a team and who work together to provide care for a panel of patients."

Inclusion Criteria:

* Primary Care Teams (PCTs) must be able to function as a single randomization unit with low risk of contamination between participants and physicians due to the absence of blinding in the intervention (see section 8.8 for details on blinding).
* PCT must have a sufficient number of patients meeting modifiable high-risk patient criteria (see section 8.1 on sample size estimates).
* PCT must express willingness to be randomized to either receive the CONQUEST program initially, or usual care until program roll-out to the delayed intervention arm.

Exclusion Criteria:

* PCTs that are in the process of, or planning to change EHR software provider or practice ownership within the trial outcome evaluation period
* PCTs engaged in active research studies or COPD related Quality Improvement Programs which might impact the ability to implement CONQUEST program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1a: COPD Exacerbations and 1b) major cardiac or respiratory events | During the 2-year outcome evaluation period
  To evaluate the effectiveness of the CONQUEST program on 1a) the annual rate of moderate or severe COPD exacerbations and on 2b) the annual rates of major adverse cardiac or respiratory events (during the outcome evaluation period).

SECONDARY OUTCOMES:
Systemic corticosteroid use (SCS) | During the 2 year outcome evaluation period
  To evaluate the impact of the CONQUEST program on systemic corticosteroid (SCS) use to treat COPD exacerbations during the outcome evaluation period.

OTHER OUTCOMES:
Exploratory Objective 1: The rate of explanatory diagnoses other than COPD | During implementation and outcome evaluation period, 2.5 years
  To evaluate the impact of the CONQUEST program on the rate of explanatory diagnoses other than COPD, diagnosed during the implementation or outcome evaluation periods.
Exploratory Objective 2: Lung function | During implementation and outcome evaluation period, 2.5 years
  To evaluate the impact of the CONQUEST program on lung function.
Exploratory Objective 3: Health status | During implementation and outcome evaluation period, 2.5 years
  To evaluate the impact of the CONQUEST program on COPD health status.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - Mount Sinai, New York, New York
  - MetroHealth, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hickman K, Tarabichi Y, Dickens AP, Pullen R, Kerr M, Couper A, Evans A, Gatenby J, Alves L, Ariti C, Bafadhel M, Carter V, Chalmers J, Chen R, Devereux G, Drummond MB, Gibson JM, Halpin DMG, Han M, Hanania NA, Hurst JR, Kaplan A, Kostikas K, Make B, Mapel D, Marshall J, Martinez F, Meldrum C, van Melle M, Miravitlles M, Morris T, Mullerova H, Murray R, Muro S, Nordon C, Ohar J, Pace W, Pollack M, Quint JK, Sharma A, Singh D, Singh M, Trudo F, Williams D, Wilkinson T, Winders T, Price D. Pragmatic Evaluation of an Improvement Program for People Living With Modifiable High-Risk COPD Versus Usual Care: Protocols for the Cluster Randomized PREVAIL Trial. Chronic Obstr Pulm Dis. 2025 May 27;12(3):223-239. doi: 10.15326/jcopdf.2024.0564. PMID 40300198